CLINICAL TRIAL: NCT01112384
Title: A Phase II Study of SB939 in Patients With Translocation-Associated Recurrent/Metastatic Sarcomas
Brief Title: A Study of SB939 in Patients With Translocation-Associated Recurrent/Metastatic Sarcomas
Acronym: IND200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I200
Record Dates: First submitted 2010-04-14; First posted 2010-04-28 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB939 (Experimental)
  Interventions: Drug: SB939

INTERVENTIONS:
Drug: SB939 — Given orally 3 times per week

SUMMARY:
The purpose of this study is to find out what effects a new drug SB939 has on you and your sarcoma.

This research is being done because there is a need for better treatment options for advanced or recurring sarcoma.

SB939 has been shown to shrink tumours in animals and some people and seems promising but it is not clear if it has any positive effects in sarcoma.

DETAILED DESCRIPTION:
Objectives:

1. - To determine the efficacy of SB939 in translocation associated sarcoma patients.
2. - To determine response duration, stable disease rate and progression free survival.
3. - To evaluate toxicity of SB939.
4. - To investigate potential molecular factors predictive of response.

60mg SB939 will be given every other day 3 times a week for 3 weeks followed by a week off. Patients may receive a maximum of 12 cycles if they have a response to treatment in the absence of disease progression or unacceptable toxicity. Patients with stable disease may continue therapy for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically diagnosed sarcomas that are associated with chromosomal translocation producing a fusion transcription factor oncogene.
* Patients must have measurable disease.
* A tissue block from primary or metastatic tumor must be available for confirmation of diagnosis, translocation subtype and correlative studies.
* Up to 1 prior chemotherapy regimen in the metastatic setting is permitted providing 28 days have elapsed.
* Prior radiation permitted provided a minimum of 28 days have elapsed.
* Surgery permitted provided at least 3 weeks have elapsed.
* Prior hormone therapy permitted.
* Patients must have life expectancy ≥ 12 weeks.
* Metastatic or locally recurrent disease incurable with standard treatment.
* Acceptable end-organ function. ECOG 0, 1 or 2.
* granulocytes ≥1.5x10/9/L
* platelets ≥100x10/9/L
* bilirubin ≤UNL
* potassium ≤UNL
* calcium, magnesium within normal limits
* AST, ALT ≤2.5 x UNL
* serum creatinine ≤UNL or creatinine clearance ≥50mL/min
* QTc ≤450m sec
* LVEF ≥50%
* Troponin I or T ≤ UNL

Exclusion Criteria:

* Cardiac exclusions; Patients with any preexisting uncontrolled cardiac condition.
* History of myocardial infarction at any time in the past.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 5 years.
* Patients with documented CNS metastases, unless adequately treated with radiation at least 30 days prior to enrollment. Patients cannot have concurrent anti-convulsants or dexamethasone for control of symptoms. Patients with leptomeningeal disease, even with treatment, cannot be enrolled due to generally poor prognosis.
* Inability to take oral medication. Patients must be able to swallow SB939 capsules and have no gastrointestinal abnormalities (e.g. bowel obstruction or previous gastric resection) which would lead to inadequate absorption of SB939.
* Previous treatment with an HDAC inhibitor.
* Treatment with another investigational therapy or other anticancer therapy within 28 days prior to study entry.
* Known HIV, hepatitis B or hepatitis C infections.
* Dysrhythmic drugs - use of agents with a known risk of Torsades De Pointe is not permitted during the study. A comprehensive list can be found at http://torsades.org.
* Presence of any chronic medical condition or comorbidity such as pulmonary disease, active CNS disease, active infection, psychiatric condition, or laboratory abnormality that may increase the risks associated with study participation/study drug administration or may interfere with the interpretation of study results.
* Women or men who are not sterile unless they use an adequate method of birth control. Female patients that are post-menopausal for at least 12 months or are surgically sterile are considered sterile.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2013-01-21 (Actual); Study Completion 2014-01-16 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy (as measured by objective response) of SB939 when given orally every other day 3 times a week, in patients with translocation-associated sarcomas. | 24 months
  The primary endpoint of this study is objective tumour response using RECIST 1.1 [Eisenhauer 2009]. Response is defined as 30% decrease in the sum of the diameters of the target lesions (partial response) maintained for at least 4 weeks, or complete disappearance of disease and cancer related symptoms (complete response), also maintained for at least 4 weeks. The median and range of the duration of response will be assessed. A 95% confidence interval for the true objective response rate will be given.

SECONDARY OUTCOMES:
Response duration, stable disease rate and progression free survival in these patients. | 24 months
Tolerability and toxicity of SB939, according to NCI CTCAE 4.0, in this population | 24 months
Potential molecular factors predictive of response in formalin fixed paraffin embedded specimens of patient sarcoma tissue | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Chu, Study Chair — Cross Cancer Institute
Locations (8):
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chu QS, Nielsen TO, Alcindor T, Gupta A, Endo M, Goytain A, Xu H, Verma S, Tozer R, Knowling M, Bramwell VB, Powers J, Seymour LK, Eisenhauer EA. A phase II study of SB939, a novel pan-histone deacetylase inhibitor, in patients with translocation-associated recurrent/metastatic sarcomas-NCIC-CTG IND 200dagger. Ann Oncol. 2015 May;26(5):973-981. doi: 10.1093/annonc/mdv033. Epub 2015 Jan 28. PMID 25632070